CLINICAL TRIAL: NCT01996683
Title: A Randomized Prospective Comparative Study of Efficacy and Safety of Continued Iron Chelation Therapy In Poly-transfused Thalassemia Patients With Low Serum Ferritin (< 500 ng/ml)
Brief Title: Efficacy and Safety of Efficacy and Safety of Continued Iron Chelation Therapy In Poly-transfused Thalassemia Patients With Low Serum Ferritin (< 500 ng/ml)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iron chelation in thalassemia
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Beta-thalassemia; Serum Ferritin; Iron Chelation Therapy
Keywords: B-thalassemia; ferritin
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferoxamine; Deferiprone; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iron chelation (Active Comparator): Included 25 thalassemia patients with low serum ferritin (< 500) or downward ferritin trend inspite of reduction of chelation dose over the last 6 months. They will continue their chelation therapy.
  Interventions: Drug: desferal, ferriprox, blood transfusion
- blood transfusion only (Placebo Comparator): Included 25 thalassemia patients with low serum ferritin (< 500) or downward ferritin trend inspite of reduction of chelation dose over the last 6 months. They will be subjected to discontinuation of their chelation therapy.
  Interventions: Drug: desferal, ferriprox, blood transfusion

INTERVENTIONS:
Drug: desferal, ferriprox, blood transfusion — Deferiprone (75-100 mg/kg/d) and deferoxamine (20-60 mg/kg/d) aimed at achieving "normal" body iron stores in poly-transfued arm1.
  Arm 2 will only recieve blood transfusion with no chelation
  Other Names: deferiprone; deferoxamine

SUMMARY:
safety and efficacy of different iron chelation therapy in transfusion dependent beta-thalaasemia patients with low serum ferritin and continued regular transfusion regimen.

DETAILED DESCRIPTION:
Treatment of transfusional iron overload in TM patients with low serum ferritin (continued decrease in serum ferritin ) even after reduction of chelation dose.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with low transfusional iron overload secondary to thalassemia major showing downward-trend in SF over last 6 months ( 2 readings are needed).

  * Thalassemia major patients with SF equal or less than 500 after reduction of chelation dose. Patients on different types of chelation monotherapy will be included
  * The subjects must also have a level of understanding and willingness to cooperate with the confinement and procedures described in the consent form and scheduled by the study site. In addition, he/she must be able to provide voluntary written informed assent or consent forms.

Exclusion Criteria:

* subjects with HIV positive or have active HCV.
* A history of serious immunologic hypersensitivity to any medication such as anaphylaxis or angioedema.
* Participation in a previous investigational drug study within the 30 days preceding screening.
* A woman of childbearing potential must have a negative serum pregnancy test at screening. She must use a medically acceptable form of birth control during the study and for a month afterwards who are pregnant or breast-feeding.
* An inability to adhere to the designated procedures and restrictions of this protocol.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
downward-trend of SF(serum ferritin) over previous 6 months after reduction of chelation dose with continuation of regular transfusion regimen. | 6 month
  non inferiority of discounting chelation compared with continuing chelation in thalassemia patients with low serum ferritin and/or showing a downward-trend of SF(serum ferritin) over previous 6 months after reduction of chelation dose with continuation of regular transfusion regimen.

SECONDARY OUTCOMES:
safety and occurrence of AEs in both studied groups (with and without chelation) in relation to different chelation therapy. | 12 month
  determine the safety and occurrence of AEs in both studied groups (with and without chelation) in relation to different chelation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen S. Elalfy, professour, Principal Investigator — Ain Shams University
Locations (1):
- Pediatric Hematology clinic, Ain Shams University, Cairo, Egypt